CLINICAL TRIAL: NCT01173276
Title: Intrauterine Insemination In HIV-Discordant Couples
Acronym: ARTEMIS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The field has changed, and we have decided to develop a PrEP program.
Sponsor: Boston Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARTEMIS
Record Dates: First submitted 2010-07-28; First posted 2010-08-02 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2012-01

CONDITIONS: HIV-1; Fertility; Infertility
Keywords: Acquired Immune Deficiency Syndrome; Assisted Reproductive Technology; Fertility; HIV; HIV Discordant; Infertility; Intrauterine Insemination; Sexually Transmitted Diseases; Sperm Washing
MeSH Terms: conditions — Infertility; Acquired Immunodeficiency Syndrome; Sexually Transmitted Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Sperm Washing with Intrauterine Insemination (IUI) — For semen samples, seminal fluid will be separated from sperm using a density gradient/swim-up separation technique. The purified sperm sample will be washed, and screened for HIV RNA using sensitive real-time RT-PCR. Samples with detectable traces of HIV RNA will not be used for insemination. Samples with no detectable traces of HIV RNA will be used for a standard intrauterine insemination of the female partner.

SUMMARY:
This study aims to assess the feasibility of a novel standard of care technique for intrauterine insemination (IUI) in HIV-discordant couples in the United States. This study will involve couples in which the male partner is HIV positive, but the female partner is negative. The investigators will institute a protocol similar to those used presently throughout Europe with good success. To date, no HIV seroconversions have occurred in over 4000 inseminations performed in HIV serodiscordant couples. All male subjects will be on stable HAART, and have undetectable serum viral loads prior to insemination. Semen samples will be subjected to a stringent sperm wash procedure and screened for HIV RNA. Female subjects will be followed post-insemination for seroconversion and pregnancy. Infants will be followed for seroconversion at birth through 4 months of age.

DETAILED DESCRIPTION:
This study aims to assess the feasibility of a novel standard of care technique for intrauterine insemination (IUI) in HIV-discordant couples in the United States. This study will involve couples in which the male partner is HIV positive, but the female partner is negative.

The investigators will institute a protocol similar to those used presently throughout Europe with good success. To date, no HIV seroconversions have occurred in over 4000 inseminations performed in HIV serodiscordant couples.

All male subjects will be on stable HAART and have undetectable serum viral loads prior to insemination. For semen samples, seminal fluid will be separated from sperm using a density gradient/swim-up separation technique. The purified sperm sample will be washed, and screened for HIV RNA using sensitive real-time RT-PCR. Samples with detectable traces of HIV RNA will not be used for insemination. Samples with no detectable traces of HIV RNA will be used for a standard intrauterine insemination of the female partner.

Female subjects will be followed post-insemination for seroconversion and pregnancy. Infants will be followed for seroconversion at birth through 3 months of age.

The data being collected in this pilot feasibility study will be mostly descriptive, lacking sample size to achieve statistical power for testing. However, the investigators will use case-control analysis to compare couples who achieve pregnancy with those who do not across demographics and markers of HIV disease progression. Additionally, the investigators have developed a 14 item, 5-point Likert scale to assesses the psychosocial impact of reproductive health issues stemming from HIV-discordance in both the female and male participants.

The expected duration for any unique subject couple is 3 to 12 months, depending on pregnancy. It is expected that the interventional portion of this study will continue for up to 2 years, depending on pregnancies.

ELIGIBILITY:
Inclusion Criteria:

* Couples with HIV discordance with an HIV seronegative female partner and HIV seropositive male partner
* Men must be HIV positive with an undetectable viral load (<75 copies/ml)
* Men must be clinical stable on antiretroviral therapy for 6 months
* Men must have a CD4 count > 250 at screening
* Men must be between 18-50 years of age
* Men must have a baseline test sperm preparation demonstrating at least 10 million motile sperm per sample
* Men must have a letter of medical clearance specific for this procedure from primary care physician stating that subject is in good health and psychologically stable
* Men must be willing to have constituent follow-up of HIV care throughout study participation
* Women must have an HIV-1/HIV-2 negative serology at screening
* Women must be between 18-40 years of age
* Women must have a body mass index (BMI) less than 30
* Women must be a non-smoker
* Women must be ovulatory (as determined by LH tracking)
* Women must have normal uterine cavity with at least one documented patent fallopian tube (as determined by hysterosalpingogram)
* Women must have adequate day 3 ovarian reserves: FSH,12 mlU/ml and estradiol<80pg/ml
* Women must have no evidence of active urogenital infection at screening
* Women must have a normal PAP smear and GC/Chlamydia at screening
* Women must have a letter of medical clearance specific to this procedure from subject's primary care physician stating that subject is in good health and psychological stable.

Exclusion Criteria:

* Subjects with untreated sexually transmitted diseases (syphilis, GC, CT)
* Men with detectable viral load (>75) at screening
* Subjects with any condition (including, but not limited to alcohol and drug use), which, in the opinion of the investigator, could compromise the subject's safety or adherence to the protocol
* Subjects with any uncontrollable medical or psychiatric condition that,in the opinion of the investigator, cannot be adequately stabilized and could be considered a contraindication to participation

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2009-09; Primary Completion 2012-09 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Pregnancy | Sixteen days after IUI
  A serum pregnancy test will be performed 16 days after IUI if menses is missed.

SECONDARY OUTCOMES:
Post-IUI HIV Infection of Female Subject | Four weeks after IUI
  The female subject will be tested for HIV by branch-DNA (b-DNA) test four weeks after each insemination.
Female Subject HIV-1/HIV-2 Serology | Three, six, nine (pregnant only) and twelve months after insemination
  If the female subject does not become pregnant, she will be tested for HIV-1/HIV-2 serology at 3 months, 6 months and 12 months after the insemination. If repeat inseminations are performed, the above-stated timeline will be followed based on the last insemination performed. If the female subject does become pregnant, she will be tested for HIV-1/HIV-2 serology at 3 months, 6 months and 9 months after the insemination, and again at 3 months postpartum.
Infant HIV-1/HIV-2 Serology | Three months of age
  For a successful birth, the infant will undergo an HIV-1/HIV-2 serology test at three months of age.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret M Sullivan, MD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Background] Anderson DJ, Politch JA. Providing fertility care to HIV-1 serodiscordant couples: a biologist's point of view. Am J Bioeth. 2003 Winter;3(1):47-9. doi: 10.1162/152651603321611980. No abstract available. PMID 12859847
- [Background] Bujan L, Hollander L, Coudert M, Gilling-Smith C, Vucetich A, Guibert J, Vernazza P, Ohl J, Weigel M, Englert Y, Semprini AE; CREAThE network. Safety and efficacy of sperm washing in HIV-1-serodiscordant couples where the male is infected: results from the European CREAThE network. AIDS. 2007 Sep 12;21(14):1909-14. doi: 10.1097/QAD.0b013e3282703879. PMID 17721098
- [Background] Bujan L, Pasquier C, Labeyrie E, Lanusse-Crousse P, Morucci M, Daudin M. Insemination with isolated and virologically tested spermatozoa is a safe way for human immunodeficiency type 1 virus-serodiscordant couples with an infected male partner to have a child. Fertil Steril. 2004 Oct;82(4):857-62. doi: 10.1016/j.fertnstert.2004.02.128. PMID 15482760
- [Background] Centers for Disease Control (CDC). Semen banking, organ and tissue transplantation, and HIV antibody testing. MMWR Morb Mortal Wkly Rep. 1988 Feb 5;37(4):57-8, 63. No abstract available. PMID 3122014
- [Background] Centers for Disease Control (CDC). HIV-1 infection and artificial insemination with processed semen. MMWR Morb Mortal Wkly Rep. 1990 Apr 20;39(15):249, 255-6. No abstract available. PMID 2109169
- [Background] Centers for Disease Control and Prevention. Revised guidelines for HIV counseling, testing, and referral. MMWR Recomm Rep. 2001 Nov 9;50(RR-19):1-57; quiz CE1-19a1-CE6-19a1. PMID 11718472
- [Background] Englert Y, Van Vooren JP, Place I, Liesnard C, Laruelle C, Delbaere A. ART in HIV-infected couples: has the time come for a change of attitude? Hum Reprod. 2001 Jul;16(7):1309-15. doi: 10.1093/humrep/16.7.1309. PMID 11425804
- [Background] Ethics Committee of the American Society for Reproductive Medicine. Human immunodeficiency virus and infertility treatment. Fertil Steril. 2002 Feb;77(2):218-22. doi: 10.1016/s0015-0282(01)03000-x. No abstract available. PMID 11821074
- [Background] Gilling-Smith C, Nicopoullos JD, Semprini AE, Frodsham LC. HIV and reproductive care--a review of current practice. BJOG. 2006 Aug;113(8):869-78. doi: 10.1111/j.1471-0528.2006.00960.x. Epub 2006 Jun 2. PMID 16753050
- [Background] Gilling-Smith C, Smith JR, Semprini AE. HIV and infertility: time to treat. There's no justification for denying treatment to parents who are HIV positive. BMJ. 2001 Mar 10;322(7286):566-7. doi: 10.1136/bmj.322.7286.566. No abstract available. PMID 11238138
- [Background] Marina S, Marina F, Alcolea R, Exposito R, Huguet J, Nadal J, Verges A. Human immunodeficiency virus type 1--serodiscordant couples can bear healthy children after undergoing intrauterine insemination. Fertil Steril. 1998 Jul;70(1):35-9. doi: 10.1016/s0015-0282(98)00102-2. PMID 9660417
- [Background] Pasquier C, Anderson D, Andreutti-Zaugg C, Baume-Berkenbosch R, Damond F, Devaux A, Englert Y, Galimand J, Gilling-Smith C, Guist'hau O, Hollander L, Leruez-Ville M, Lesage B, Maillard A, Marcelin AG, Schmitt MP, Semprini A, Vourliotis M, Xu C, Bujan L; CREAThE Network. Multicenter quality control of the detection of HIV-1 genome in semen before medically assisted procreation. J Med Virol. 2006 Jul;78(7):877-82. doi: 10.1002/jmv.20636. PMID 16721844
- [Background] Politch JA, Xu C, Tucker L, Anderson DJ. Separation of human immunodeficiency virus type 1 from motile sperm by the double tube gradient method versus other methods. Fertil Steril. 2004 Feb;81(2):440-7. doi: 10.1016/j.fertnstert.2003.06.028. PMID 14967387
- [Background] Sauer MV. Sperm washing techniques address the fertility needs of HIV-seropositive men: a clinical review. Reprod Biomed Online. 2005 Jan;10(1):135-40. doi: 10.1016/s1472-6483(10)60815-2. PMID 15705311
- [Background] Sauer MV, Wang JG, Douglas NC, Nakhuda GS, Vardhana P, Jovanovic V, Guarnaccia MM. Providing fertility care to men seropositive for human immunodeficiency virus: reviewing 10 years of experience and 420 consecutive cycles of in vitro fertilization and intracytoplasmic sperm injection. Fertil Steril. 2009 Jun;91(6):2455-60. doi: 10.1016/j.fertnstert.2008.04.013. Epub 2008 Jun 13. PMID 18555235
- [Background] Semprini AE, Bujan L, Englert Y, Smith CG, Guibert J, Hollander L, Ohl J, Vernazza P. Establishing the safety profile of sperm washing followed by ART for the treatment of HIV discordant couples wishing to conceive. Hum Reprod. 2007 Oct;22(10):2793-4; author reply 2794-5. doi: 10.1093/humrep/dem197. Epub 2007 Jul 3. No abstract available. PMID 17609245